CLINICAL TRIAL: NCT01620450
Title: A Single-centre, Randomised, Double Blind, Cross-over Trial Demonstrating the Bioequivalence Between NN2000-Mix30 and NN-X14Mix30 (NovoRapid® 30 Mix) in Healthy Japanese Subjects
Brief Title: Comparison of Insulin Aspart Produced by Current Process and the NN2000 Process in Healthy Japanese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2000-1612
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — biphasic human insulin 30

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NN2000 (Experimental)
  Interventions: Drug: biphasic human insulin 30
- NN-X14 (Active Comparator)
  Interventions: Drug: biphasic human insulin 30

INTERVENTIONS:
Drug: biphasic human insulin 30 — Single dose of each formulation administered subcutaneously (s.c., under the skin) on two separate visits

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to compare insulin aspart produced by current process and the NN2000 process in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese
* Considered generally healthy based on medical history and physical examination
* Body Mass Index (BMI) between 18 and 27 kg/m^2 (both inclusive)
* Fasting plasma glucose between 3.8 mmol/L (68.4 mg/dL) and 6.0 mmol/L (108.0 mg/dL)

Exclusion Criteria:

* Clinically significant abnormal values in clinical laboratory tests of haematology, biochemistry, fasting plasma glucose and urinalysis
* Any serious systemic infectious disease that occurred during the last 4 weeks before trial
* Any inter-current illness that may affect blood glucose
* Subject with a first degree relative with diabetes mellitus
* Blood donation of more than 400 mL (inclusive) in total within the last 12 weeks or more than 200 mL (inclusive) in total within the last 4 weeks

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2004-11-20 (Actual); Primary Completion 2005-02-26 (Actual); Study Completion 2005-02-26 (Actual)

PRIMARY OUTCOMES:
Area under the curve of insulin aspart concentration (AUC IAsp, 0-16h) | From 0 to 16 hours after injection
Maximum insulin aspart concentration (Cmax IAsp)

SECONDARY OUTCOMES:
Area under the curve of insulin aspart concentration (AUC IAsp)
Time to maximum insulin aspart concentration (tmax IAsp)
Terminal elimination half life (t½)
Body weight
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com